CLINICAL TRIAL: NCT06568991
Title: The Effect of Low-protein Rice on Nutritional Status and Other Outcomes of Patients With Chronic Kidney Disease.
Brief Title: The Effect of Low-protein Rice on Nutritional Status and Other Outcomes of Patients With Chronic Kidney Disease.(KS01)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Collaborators: TAIWAN KITOKU CO., LTD. (Unknown)
Responsible Party: Principal Investigator, Shang-Jyh,Hwang, Associate Dean, Kaohsiung Medical University Chung-Ho Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KMUHIRB-F(II)-20150030
Record Dates: First submitted 2022-02-09; First posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Chronic Kidney Disease (CKD)
Keywords: low protein; chronic kidney disease; nutritional
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Observational control group (Placebo Comparator): Giving a meal plan and nutrition education. It need to define recruited subject intake low-protein formula's frequency ≦ 3 times/week
  Interventions: Dietary Supplement: Low Protein Rice MATSUBUMAI
- the True Low Protein Rice group (Active Comparator): Use low protein rice to replace staple food in two meals during a day.
  Interventions: Dietary Supplement: Low Protein Rice MATSUBUMAI

INTERVENTIONS:
Dietary Supplement: Low Protein Rice MATSUBUMAI — Investigators will recruit 100 subjects participating in the"PRE-ESRD education plan" at KMUH. Subjects will receive dietary education of low protein diet (providing energy 25 to 35 Kcal/Kg/day, protein 0.6 to 0.8 g/Kg/day) by dietitians. Subjects will be randomly assigned to a observational group or rue low protein rice group.

SUMMARY:
1. To examine nutrient intake change in chronic kidney disease patients consuming " Low Protein Rice MATSUBUMAI "compared to a regular care group at 0,1,3,6 month.
2. To assess nutritional status improved or maintained after low protein rice intervention.
3. To assess whether the patient's renal function improved or maintained after low protein rice intervention.

DETAILED DESCRIPTION:
1. Recruited the subjects procedures A physical checking the history and blood biochemical data will be carried out by the study physician to verify eligibility for enrollment study at outpatient. A physical explain and answer about the study procedure and criteria to subjects.

   Subjects review informed consent and sign it.
2. The trail procedures(brief describe)

1.After the subjects will sign informed consent form at the outpatient, they will be enrolled (phone) and schedule study visit1 (M0) by study staff. 2.The study visit1 will collect demographics, blood, urine and distribute product and product consumption diaries, and perform SGA (Subjective Global Assessment). 3.The study visit2 (M1), after the product be used for 4 weeks, will collect adverse event, blood,urine, and SGA. 4.The study visit3(M3), after the product be used for 12 weeks, will collect adverse event, blood,urine, and SGA. 5.The study visit4(M6), after the product be used for 24 weeks, will collect adverse event, blood,urine, and SGA. 3.Subject and study design： Investigators will recruit 100 subjects participating in the"PRE-ESRD education plan" at KMUH.

Subjects will receive dietary education of low protein diet (providing energy 25 to 35 Kcal/Kg/day, protein 0.6 to 0.8 g/Kg/day) by dietitians. Subjects will be randomly assigned to a observational group or rue low protein rice group. Observational group (n=40): Forty subjects will be enrolled. Subjects will receive routine dietary education of low protein diet. True Low Protein Rice group (n=60): Subjects will replace regular staple foods with low protein rice. Subjects will replace regular staple foods with low protein rice at levels of 40-160grams/ day. According to subjects' intake, subjects will be further divided into low & high intake groups for analysis. High intake group: Subjects consuming low Protein Rice at levels of 81-160 grams/day. Low intake group: Subjects consuming low Protein Rice at levels of 40-80 grams/day.

ELIGIBILITY:
Exclusion criterias

1. were undergoing dialysis
2. had cancer under any treatmen
3. had any major surgery before or after the study period
4. were pregnant or breastfeeding
5. were diagnosed with alcoholism
6. had liver, gastrointestinal tract, or other metabolic diseases
7. and/or had been determined by a physician to be clinically unstable.
8. Subject is participating in another study that has not been approved as a concomitant study by Low Protein Rice.
9. Subjects consuming oral nutritional supplement(ONS) >3 times/week for the control group and subjects consuming any ONS for the low protein rice group.

Inclusion criteria

1. Patients were diagnosed with stages 3b-5 CKD with an estimated glomerular filtration rate (eGFR) of 15-44 mL/min/1.73 m2.
2. Patients were aged 30-70 years
3. Patients received pre-end-stage renal disease (pre-ESRD) care under a pay-for-performance program (P4P) at the Department of Nephrology at Kaohsiung Medical University Hospital.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2015-05-26 (Actual); Primary Completion 2019-01-11 (Actual); Study Completion 2019-01-11 (Actual)

PRIMARY OUTCOMES:
albumin (g/dL) | baseline, 6 month
  nutritional indicators
nitrogen balance (g/day) | baseline, 6 month
  nutritional indicators
handgrip strength (kg) | baseline, 6 month
  nutritional indicators
blood urea nitrogen (mg/dL) | baseline, 6 month
  residual renal function
creatinine (mg/dL) | baseline, 6 month
  residual renal function
estimated glomerular filtration rate (eGFR) (mL/min/1.73m2) | baseline, 6 month
  residual renal function

SECONDARY OUTCOMES:
Body weight (kg) | baseline, 6 month
  Body composition
muscle mass (kg) | baseline, 6 month
  Body composition
fat mass (%) | baseline, 6 month
  Body composition
energy intake (Kcal/day) | baseline, 6 month
  Nutrient intakes
protein intake (g/day) | baseline, 6 month
  Nutrient intakes
potassium (mmol/L) | baseline, 6 month
  electrolytes
phosphorus (mg/dL) | baseline, 6 month
  electrolytes